CLINICAL TRIAL: NCT06849375
Title: Corneal Endothelial Assessment After Posterior Chamber Phakic Intraocular Lens Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Mahmoud Abdelhameed, Resident of ophthalmology department, Sohag University Hospitals, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med--25-1-11MS
Record Dates: First submitted 2025-02-07; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Corneal Endothelial Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- group who implant phakic IOL (Other): specular microscopy examination to assess the endothelial cells before and after phakic IOL implantation
  Interventions: Procedure: phakic IOL implantation

INTERVENTIONS:
Procedure: phakic IOL implantation — specular microscopy examination to assess endothelial cells before and after phakic IOL implantation

SUMMARY:
our primary aim of the work to assess the effect of phakic IOL implantation on corneal endothelium. we also used the specular microscope to assess the corneal endothelium

ELIGIBILITY:
Inclusion Criteria:

* Our inclusion criteria include: adults 18-35 years of age, myopia ˃ 6 D , anterior chamber depth (ACD) 2.85 mm or greater , an endothelial cell count of ≥ 2000 cells/mm2 and stable refractive history within 0.5 diopter for 1 year.

Exclusion Criteria:

* anterior chamber depth from endothelium < 2.85 mm, previous or current systemic or eye disease , surgery or trauma, pregnancy and nursing.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
corneal endothelial cells assessment | 1 year
  specular micrioscopy examination before and after phakic IOL implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Sohag Governorate, Egypt

REFERENCES:
- [Background] Reinstein DZ, MacGregor C, Archer TJ, Gupta R, Potter JG. A review of posterior chamber phakic intraocular lenses. Curr Opin Ophthalmol. 2024 Mar 1;35(2):138-146. doi: 10.1097/ICU.0000000000001018. Epub 2023 Dec 6. PMID 38059758
- [Background] Taneri S, Dick HB. Initial clinical outcomes of two different phakic posterior chamber IOLs for the correction of myopia and myopic astigmatism. Graefes Arch Clin Exp Ophthalmol. 2022 May;260(5):1763-1772. doi: 10.1007/s00417-021-05465-w. Epub 2021 Nov 6. PMID 34741659
- [Background] Chaurasia S, Vanathi M. Specular microscopy in clinical practice. Indian J Ophthalmol. 2021 Mar;69(3):517-524. doi: 10.4103/ijo.IJO_574_20. PMID 33595465
- [Background] Sridhar MS. Anatomy of cornea and ocular surface. Indian J Ophthalmol. 2018 Feb;66(2):190-194. doi: 10.4103/ijo.IJO_646_17. PMID 29380756
- [Background] DelMonte DW, Kim T. Anatomy and physiology of the cornea. J Cataract Refract Surg. 2011 Mar;37(3):588-98. doi: 10.1016/j.jcrs.2010.12.037. PMID 21333881